CLINICAL TRIAL: NCT04465344
Title: Multicentric Clinical Study to Determine Safety and Efficacy of a Hydrophobic Acrylic Trifocal Intraocular Lens (IOL)
Brief Title: Multicentric Clinical Study on Isatis TF Trifocal Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutting Edge SAS (Industry)
Collaborators: targomedGmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE2001
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-09

CONDITIONS: Cataract; Lens Opacities
Keywords: Intraocular Lens; IOL; hydrophobic; trifocal
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL implantation experimental (Experimental): Experimental arm: Trifocal intraocular lens Isatis TF
  Interventions: Device: Implantation of trifocal IOL, Isatis TF (device under investigation)
- IOL implantation active comparator (Active Comparator): Comparator arm: Monofocal intraocular lens Isatis
  Interventions: Device: Implantation of monofocal IOL, Isatis (control device)

INTERVENTIONS:
Device: Implantation of trifocal IOL, Isatis TF (device under investigation) — Patients will be implanted with study IOL in both eyes
  Arms: IOL implantation experimental
Device: Implantation of monofocal IOL, Isatis (control device) — Patients will be implanted with Control IOL in both eyes
  Arms: IOL implantation active comparator

SUMMARY:
The study will be a multicentric, prospective open-label ethics committee approved clinical study to investigate safety, visual outcomes, contrast sensitivity and rotational stability after bilateral implantation of Isatis TF IOL following cataract surgery.

DETAILED DESCRIPTION:
This is a staged, multicentric, controlled, prospective, open-label clinical study whereby patients undergoing routine cataract surgery will have bilateral implantation of hydrophobic acrylic refractive trifocal intraocular lenses (Isatis TF) or the monofocal control device Isatis.

The investigational device, Control lens and all study products, including the devices used for the study examinations, will be used within the intended use specifications from the manufacturer. In addition, no invasive or other burdening examinations will occur for the patient.

The study will be carried out in up to five clinical centers in Spain.

The device under investigation is a hydrophobic acrylic trifocal intraocular lens (IOL) manufactured by the sponsor of this study. The trifocality of this investigational device is based on a purely refractive principle with the goal to provide additional near and intermediate visual acuity with low photic side effects. The IOLs will be implanted in the course of routine cataract surgery and will benefit to patients suffering from cataract development.

The control device (Isatis) is a hydrophobic acrylic monofocal intraocular lens to be implanted during cataract surgery. This control lens is CE approved and commercially available in Spain. Isatis monofocal lens is the parent lens of the device under investigation and both lenses share mechanical and material properties.

In total 180 patients will be recruited for this clinical study and undergo bilateral implantation of the Isatis TF intraocular lens or Isatis lens in a 2:1 ratio. Subjects participating in the trial will attend a total of maximum 11 study visits over a period of 11-13 months. Subjects would have the option for unscheduled visits if required medically.

Data analyses will be performed after the last patient finished the 120-180 days postoperative examination.

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented age-related cataract in both eyes with no comorbidity;
* Calculated IOL power is within the range of the investigational IOLs;
* Male or female adults ages 50 years or older on the day of screening who have cataracts in both eyes;
* Regular corneal astigmatism (measured by topographer)
* Astigmatism ≤1.0 D (measured by an automatic keratometer)
* Clear intraocular media other than cataract;
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures;
* Patient is willing to receive bilateral implantation of a trifocal IOL (this inclusion criteria applies only to the study group, not the control group);
* Signed informed consent.

Exclusion Criteria:

* Age of patient < 50 years;
* Regular corneal astigmatism >1.0 dioptres (measured by an automatic keratometer)
* Irregular astigmatism (measured by topographer);
* Difficulty for cooperation (distance from their home, general health conditions);
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders);
* Subjects with AMD suspicious eyes as determined by OCT examination;
* Previous intraocular or corneal surgery;
* Traumatic cataract;
* Instability of keratometry or biometry measurements; Acceptable maximum standard deviation: AL: ± 150 µm; ACD: ± 150 µm; K1 / K2: ± 0.15 D;
* Ocular hypertension, suspicious glaucoma or glaucoma;
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic / scotopic conditions);
* Expected complicated surgery;
* Ocular surface disease (clinical symptoms or keratitis);
* Pregnancy or lactation;
* Second eye treatment will only be performed when Best Corrected Distance Visual Acuity (CDVA) of first eye is ≤ 0.2 logMAR (≥ 0.63 decimal);
* Concurrent participation in another drug or device investigation.

In addition to above mentioned in- and exclusion criteria, subjects shall be discontinued when certain conditions are present at the time of surgery, including:

* zonular instability;
* need for iris manipulation;
* capsular fibrosis or other opacity; and
* inability to fixate IOL in desired position. In such cases, the subject shall be followed until the condition has stabilized.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Rates of Adverse Events | 120-180 days postoperative
  The objective is to compare the SPE (Safety and Performance Endpoints) rates of the investigational product to reference data stated in the according ISO standard for posterior intraocular lenses (EN ISO 11979-7:2018) based on minimum 100 subjects.
Primary Performance Endpoint: Best Corrected Distance Visual Acuity | 120-180 days postoperative
  The primary performance endpoint is to show non inferiority of Isatis TF compared to the monofocal comparator in terms of best corrected distance visual acuity (CDVA) by means of statistical significance.

SECONDARY OUTCOMES:
Secondary Safety Endpoint: Best Corrected Distance Visual Acuity compared to historical data | 120-180 days postoperative
  The objective is to compare best corrected distance visual acuities (CDVA) above defined thresholds of the investigational product to the normative data stated in the according ISO norm (EN ISO 11979-7:2018) for posterior chamber intraocular lenses.
Secondary Performance Endpoint: Distance Corrected Near Visual Acuity (DCNVA) | 120-180 days postoperative
  Secondary performance endpoint is to show a statistically significant increase between pre-and postoperative findings on monocular Distance Corrected Near Visual Acuity (DCNVA) under photopic light conditions on the first implanted eye.
Secondary Performance Endpoint: Distance Corrected Intermediate Visual Acuity (DCIVA) | 120-180 days postoperative
  Secondary performance endpoint is to show a statistically significant increase between pre-and postoperative findings on monocular Distance Corrected Intermediate Visual Acuity (DCIVA) under photopic light conditions on the first implanted eye.

OTHER OUTCOMES:
Monocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | Preoperative, 1-2 days postoperative; 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Monocular UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Distance Visual Acuity (UDVA) under photopic light conditions | 120-180 days postoperative, 330-420 days postoperative
  Binocular UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | Preoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  Monocular CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Monocular Corrected Distance Visual Acuity (CDVA) under mesopic light conditions | 120-180 days postoperative
  Monocular CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done binocularly under mesopic light conditions.
Binocular Corrected Distance Visual Acuity (CDVA) under photopic light conditions | 120-180 days postoperative
  Binocular CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Uncorrected Intermediate Visual Acuity (UIVA) under photopic light conditions | 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Monocular UIVA is measured with ETDRS charts placed in 66cm distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Intermediate Visual Acuity (UIVA) under photopic light conditions | 120-180 days postoperative, 330-420 days postoperative
  Binocular UIVA is measured with ETDRS charts placed in 66cm distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Uncorrected Near Visual Acuity (UNVA) under photopic light conditions | 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Monocular UNVA is measured with ETDRS charts placed in 40cm distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Binocular Uncorrected Near Visual Acuity (UNVA) under photopic light conditions | 120-180 days postoperative, 330-420 days postoperative
  Binocular UNVA is measured with ETDRS charts placed in 40cm distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) under photopic light conditions | Preoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Monocular DCIVA is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) under mesopic light conditions | 120-180 days postoperative
  Monocular DCIVA is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under mesopic light conditions.
Binocular Distance Corrected Intermediate Visual Acuity (DCIVA) under photopic light conditions | 120-180 days postoperative
  Binocular DCIVA is measured with ETDRS charts placed in 66cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Monocular Distance Corrected Near Visual Acuity (DCNVA) under photopic light conditions | Preoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  Monocular DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done monocularly under photopic light conditions.
Monocular Distance Corrected Near Visual Acuity (DCNVA) under mesopic light conditions | 120-180 days postoperative
  Monocular DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under mesopic light conditions.
Binocular Distance Corrected Near Visual Acuity (DCNVA) under photopic light conditions | 120-180 days postoperative
  Binocular DCNVA is measured with ETDRS charts placed in 40cm distance with corrective glasses for far distance according to ISO 11979-7:2018. This assessment is done binocularly under photopic light conditions.
Manifest refraction | Preoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The manifest refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2018. This data will also be used to calculate the manifest refractive spherical equivalent (MRSE)
Adjusted Mean Refractive Spherical Equivalent (MRSE) | 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The predictability of the postoperative manifest refraction will be evaluated using the absolute value of the adjusted MRSE calculated by the following formula:
  MRSEadjusted = MRSEpostop - MRSEtarget.
Binocular Defocus Curve | 120-180 days postoperative
  To assess the visual acuity for different distances, defocus curves under photopic light conditions are measured. This test is performed with best distance corrected refraction and spherical additions ranging from -4.5 D to +2.0 D in 0.5 D steps. This examination is performed binocularly.
Binocular Contrast Sensitivity under photopic light conditions | 120-180 days postoperative
  Contrast Sensitivity under photopic light conditions using the standardized contrast sensitivity device CSV-1000 (VectorVision). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions | 120-180 days postoperative
  Contrast Sensitivity under mesopic light conditions using the standardized contrast sensitivity device CSV-1000 (VectorVision). This examination is performed binocularly.
Binocular Contrast Sensitivity under photopic light conditions and using a glare source | 120-180 days postoperative
  Contrast Sensitivity under photopic light conditions with a glare source using the standardized contrast sensitivity device CSV-1000 (VectorVision). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions and using a glare source | 120-180 days postoperative
  Contrast Sensitivity under mesopic light conditions with a glare source using the standardized contrast sensitivity device CSV-1000 (VectorVision). This examination is performed binocularly.
Patient reported outcomes - Quality of Vision questionnaire [McAlinden et al, 2010] | preoperative, 120-180 days postoperative
  To assess the subjective perception of disturbances by photic phenomena, the validated and verified Quality of Vision (QoV) questionnaire will be used.
  This questionnaire is a linear-scaled 30-item instrument and is designed with 10 symptoms rated in each of three scales (frequency, severity, and bothersome).
  The QoV Questionnaire provides a QoV score in terms of symptom frequency, severity, and bothersome [McAlinden et al, 2010].
Patient reported outcomes - Catquest-9SF 2011 questionnaire [Lundström et al, 2009] | preoperative, 120-180 days postoperative
  To assess if difficulties in daily life occur due to impaired sight. This questionnaire is a 9-item Rasch-scaled instrument to assess subjective perception of visual impairment after surgery [Lundström et al, 2009].
Patient reported outcomes - Patient-Reported Spectacle Independence Questionnaire (PRSIQ) [Morlock et al, 2017] | preoperative, 120-180 days postoperative
  The PRSIQ is a patient-reported measure assessing spectacle independence following cataract surgery. The analyses conducted provide evidence for the use of the PRSIQ total score as a measure of spectacle independence [Morlock et al, 2017].
Pupil Size under photopic light conditions | preoperative, 120-180 days postoperative
  Photopic pupil diameters are measured with a ruler allowing for a precision of at least +/-0.5 mm. In addition to the measurement with a ruler, pupil diameters under photopic light conditions will be recorded from the preoperative Pentacam measurement.
  For the photopic pupil diameters, eye illumination should be identical to that used for photopic contrast sensitivity testing. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 5 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Pupil Size under mesopic light conditions | preoperative, 120-180 days postoperative
  Mesopic pupil diameters are measured with a ruler allowing for a precision of at least +/-0.5 mm. For the mesopic pupil diameters, eye illumination should be identical to that used for mesopic contrast sensitivity testing. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 5 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus examination with dilated pupil | preoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination - Corneal status | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Slitlamp examination - Iris status | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Iris Status
Slitlamp examination - Signs of inflammation | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  * Signs of inflammation
  * Anterior chamber cells,
  * Anterior chamber flare,
  * Cystoid macular oedema,
  * Hypopyon, and
  * Endophthalmitis.
Slitlamp examination - Pupillary block | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Pupillary block.
Slitlamp examination - Retinal detachment | preoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Retinal detachment.
Slitlamp examination - Status of anterior and posterior capsule | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - Status of anterior and posterior capsule.
Slitlamp examination - IOL decentration | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL decentration.
Slitlamp examination - IOL tilt | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL tilt.
Slitlamp examination - IOL discoloration | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL discoloration.
Slitlamp examination - IOL opacity | 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  - IOL opacity.
Intraocular pressure (IOP) measurement | Preoperative, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative, 330-420 days postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Keratometry | Preoperative
  Keratometric measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
IOL power and target refraction | day of surgery
  The parameter of the implanted IOL must be recorded as well as the target refraction given by the IOL calculator. This parameter is needed to calculate the accuracy of achieving the target refraction. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus OCT | Preoperative
  An OCT (optical coherence tomography) image will be taken at the preoperative visit to identify AMD suspicious eyes that need to be excluded from this study. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Biometry | Preoperative
  Biometry measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Corneal topography | Preoperative
  Pentacam device (Oculus, Germany) will be used to perform corneal topography. This examination is needed to exclude patients showing an irregular corneal astigmatism.
Corneal aberrometry | Preoperative
  Pentacam device (Oculus, Germany) will be used to perform corneal aberrometry measurement. The following values will be evaluated in this study: Spherical aberrations, high order aberrations.
IOL rotation | day of surgery, 1-2 days postoperative, 7-14 days postoperative, 30-60 days postoperative, 120-180 days postoperative
  To determine the rotational stability of the lenses after implantation, the actual IOL orientation has to be recorded as the intended surgical position during surgery using a photograph through the surgery microscope or within one hour after surgery using a photograph through a slit lamp to document the rotational position of the IOL. Additional orientations are measured and recorded at the follow up visits by taking retroilluminated photographs in mydriasis using the slit lamp.
  To determine the rotational stability, it is important that the IOL axis marks of the IOL are visible as well as concurrent structures of the eye (in the same image) that are fixed and stable. Preferred fixed structures are limbal vessels. The pupil is dilated if necessary to visualize the IOL axis marks.
Halo and glare scores | Preoperative, 120-180 days postoperative, 330-420 days postoperative
  A Halo and Glare simulator software (Eyeland Design Network GmbH, Germany) will be used to assess the subjective perception of photic phenomena. The patients will be asked to adjust the halo and glare level in a simulated image to the amount they perceive of such photic phenomena. This test is performed pre- and postoperatively. The preoperative outcomes serve as a baseline measurement.

CONTACTS AND LOCATIONS:
Locations (7):
- Czechia (3):
  - Gemini Eye Clinic Ostrava, Ostrava
  - Gemini Eye Clinic Praha-Krc, Prague
  - Gemini Eye Clinic Zlín, Zlín
- Spain (4):
  - Hospital Donostia, Donostia / San Sebastian
  - Oftalvist Madrid, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205
- [Background] Morlock R, Wirth RJ, Tally SR, Garufis C, Heichel CWD. Patient-Reported Spectacle Independence Questionnaire (PRSIQ): Development and Validation. Am J Ophthalmol. 2017 Jun;178:101-114. doi: 10.1016/j.ajo.2017.03.018. Epub 2017 Mar 22. PMID 28341605
- [Background] Lundstrom M, Pesudovs K. Catquest-9SF patient outcomes questionnaire: nine-item short-form Rasch-scaled revision of the Catquest questionnaire. J Cataract Refract Surg. 2009 Mar;35(3):504-13. doi: 10.1016/j.jcrs.2008.11.038. PMID 19251145